CLINICAL TRIAL: NCT05539534
Title: Effect of Suicide Prevention Training for Professionals on Knowledge and Attitudes Regarding Suicide Prevention
Brief Title: Effect of Suicide Prevention Training for Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018/1329
Record Dates: First submitted 2021-11-29; First posted 2022-09-14 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): This is a one-arm trial. The intervention group receives a training on suicide prevention.
  Interventions: Behavioral: Training on suicide prevention

INTERVENTIONS:
Behavioral: Training on suicide prevention — Suicide prevention training in Flanders is organised by the Centre for the Prevention of Suicide and the suicide prevention workers of the Centra for Mental Health Care. These trainings are announced via the website zelfmoord1813.be/vormingen or are organized on demand. When a participant registers, they will be invited to participate in the study one week before the training.

SUMMARY:
Annually a substantial number of courses and trainings are organised in Flanders with regard to suicide prevention.These trainings are mainly aimed at intermediaries, such as caregivers, teachers, police, etc. From previous research it appears that such trainings are one of the most effective strategies for increasing knowledge, attitudes, skills and self-confidence with regard to dealing with persons who are suicidal and with crisis situations. However, such research has not yet been conducted in Flanders, which means that the effect of the training on the knowledge and attitudes of the intermediaries could not yet be determined. Therefore, this study aims to determine the effect of the trainings in Flanders. These trainings are organised by the Centre for the Prevention of Suicide (CPZ) and by the suicide prevention workers of the Centers for Mental Health Care.

All participants who register for one of these trainings will be invited by e-mail at three moments to complete an online questionnaire:

* Pre-test: one week before the training,
* Post-test: after the training,
* Follow-up: three months after training.

ELIGIBILITY:
Inclusion Criteria:

* Participating in a suicide prevention training organised by 'Centrum ter Preventie van Zelfdoding' or 'Suïcidepreventiewerking Centra Geestelijke Gezondheidszorg'

Exclusion Criteria:

* Not participating in a suicide prevention training organised by 'Centrum ter Preventie van Zelfdoding' or 'Suïcidepreventiewerking Centra Geestelijke Gezondheidszorg'

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of knowledge and attitudes on suicide and suicide prevention | Change in knowledge and attitudes at baseline (i.e., from one week before the start of the training) compared to post-test (immediately after the training, i.e. up to 3 days) and follow-up (3 months after post-test)
  Self-developed questionnaire about knowledge and attitudes on suicide and suicide prevention based on the Attitudes about Suicide Scale (ATTS).

SECONDARY OUTCOMES:
Rate of responses to suicide | Change in Response to suicide at baseline (i.e., from one week before the start of the training) compared to post-test (immediately after the training, i.e. up to 3 days) and follow-up (3 months after post-test)
  ONLY APPLICABLE FOR TRAININGS THAT LAST MORE THAN 3 HOURS. Questionnaire Responses to Suicide is a Dutch questionnaire (original name: Vragenlijst Reacties op Suïcidaliteit (VROS). This questionnaire assesses how appropriately someone can react to suicide. The lower the score, the better the person knows how to react.

OTHER OUTCOMES:
Socio-demographic characteristics | Baseline (i.e., from one week before the start of the training)
  Socio-demographic characteristics such as gender, age, and work.
Evaluation of the training | Post-test (immediately after the training, i.e. up to 3 days)
  Self-developed questionnaire about how the participants experienced the training, i.e. how satisfied they were, how applicable the training was, and an overall score of the training.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided